CLINICAL TRIAL: NCT01553825
Title: Assessment of Patient Experience During Treatment for Cancer
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-22490; SU-03082012-9290 (Other: Stanford University); VAR0075 (Other: OnCore); IRB-22490 (Other: Stanford IRB)
Record Dates: First submitted 2012-03-12; First posted 2012-03-14 (Estimated); Last update posted 2020-04-29 (Actual); Status verified 2019-04

CONDITIONS: Carcinoma
MeSH Terms: conditions — Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pathologically diagnosed carcinoma

SUMMARY:
Assessing the mindset of cancer patients will help us better understand which patients are having difficulty dealing with the diagnosis and treatment that may not otherwise be fully appreciated by their physicians. By identifying such patients, we may then be able to design and implement strategies that can help improve their coping skills both during the treatment as well as after the completion of treatment. In addition to addressing physical concerns and symptoms, this approach will help address the overall emotional impact of a cancer diagnosis as more patients are living as cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically diagnosed carcinoma patients at Stanford cancer center who signed the informed consent form.

Exclusion Criteria:

* Patients with a prognosis of < 6 months life expectancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pathologically diagnosed carcinoma patients at Stanford cancer center who signed the informed consent form.
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Horst, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States